CLINICAL TRIAL: NCT06300060
Title: The Effect of a Synbiotic Formulation on Endurance Exercise Performance in Trained Cyclists: A Randomized, Double-Blinded, Placebo-Controlled, Parallel Trial
Brief Title: Synbiotic Supplementation in Cyclists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Principal Investigator, Dr. Raylene Reimer, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: REB23-1161
Record Dates: First submitted 2024-02-26; First posted 2024-03-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Exercise Endurance
Keywords: Exercise; Cyclists; Athlete; Synbiotic; Prebiotic; Probiotic; Gut microbiota; Metabolism
MeSH Terms: conditions — Motor Activity | interventions — Synbiotics

STUDY DESIGN:
Intervention Model Description: Parallel arm. Single-site, double-blinded, placebo-controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The synbiotic and placebo are both powders identical in taste and appearance and are equally dissolvable in cold water.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic (Experimental): Participants receive the synbiotic for 6 weeks.
  Interventions: Dietary Supplement: Synbiotic
- Placebo (Placebo Comparator): Participants receive the placebo for 6 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic — Combination of a probiotic and prebiotic. Daily administration in a single dose in powder form.
  Arms: Synbiotic
Dietary Supplement: Placebo — Placebo. Daily administration in a single dose in powder form.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the efficacy of a synbiotic blend on exercise performance and other exercise parameters in trained adult cyclists. It is hypothesized that those taking the synbiotic blend will have improved endurance exercise performance.

The primary objective is to assess the impact of a synbiotic on 20km distance trial performance in 36 cyclists. Secondary objectives include assessing the impact of the synbiotic on exercise metabolism, body composition, gastrointestinal and immune health.

DETAILED DESCRIPTION:
The goal of this randomized double-blinded clinical trial is to evaluate the potential beneficial effects of a synbiotic formulation on exercise performance in trained adult cyclists. The main questions it aims to answer are related to the Synbiotic effects on:

* Cycling performance
* Exercise metabolism
* Gastrointestinal health
* Immune system
* Body composition
* Fecal Short Chain Fatty Acids (SCFAs)
* Fecal microbiome composition

Participants will be recruited and, if consenting and eligible, will undergo the initial pre-testing phase for baseline assessment (4 on-site visits). Then, they will be randomized to receive the synbiotic or placebo and instructed to consume one sachet daily for 42 consecutive days. After 4-5 weeks of intervention (Day 33), post-testing phase will start, and participants will be asked to return to the site to perform post testing assessments (over 4 on-site visits). Study visits will occur as follows, V1 (Day -9), V2 (Day -6), V3 (Day -3), V4 (Day 0), V5 (Day 33), V6 (Day 36), V7 (Day 39), and V8 (Day 42).

Researchers will compare the assessed outcomes to baseline in each group and evaluate the difference between groups following the synbiotic consumption to highlight any statistically and clinically relevant observations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18-45
* Currently cycling for at least 3 hours per week for the past 3 months
* Free of any contraindications to exercise and any medical condition that could interfere with or influence metabolic or cardiovascular responses to exercise
* Have a resting heart rate <100 bpm and resting systolic and diastolic blood pressures <160 mmHg and <90 mmHg, respectively.

Exclusion Criteria:

* Use of antibiotics or probiotic products within 4 weeks prior to study enrollment (note: participants will be eligible after a 2-week washout period)
* Current laxative use
* Are a smoker or use tobacco products
* Consume >21 units of alcohol per week
* Have donated blood in the previous 3 months
* Have a BMI ≥30kg/m2
* Are pregnant or lactating or planning to become pregnant for the duration of the study
* Are dieting for weight loss or are following a low carbohydrate diet
* Have participated in another clinical trial within the 30 days preceding study enrollment
* Are taking medications known to affect cardiovascular or metabolic responses to exercise
* Have a medical condition that could interfere with study intervention and assessment
* Have current musculoskeletal injuries that limit exercise capacity
* Are non-English speaking

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Change in endurance exercise performance measured during a 20km cycling distance trial | 42 Days
  Assessed as time (minutes) to complete 20km cycling distance

SECONDARY OUTCOMES:
Change in maximal oxygen consumption (V̇O2max) measured during a Step-Ramp-Step Test | 36 Days
  Assessed as mL·kg-1·min-1 measured through expired air collection
Change in peak power output (PPO) measured during a Step-Ramp-Step Test | 36 Days
  Assessed as highest power output in Watts
Change in power output corresponding to the gas exchange threshold (GET) and respiratory compensation point (RCP) | 36 Days
  Assessed as power output in Watts at GET and RCP
Change in time to exhaustion measured during a cycling session at 85% of the peak power output | 39 Days
  Assessed as time (minutes) to reach volitional exhaustion.
Change in fat and carbohydrate oxidation measured during exercise sessions | 36, 39 and 42 Days
  Assessed with the nonprotein respiratory quotient equation using expired air variables (VO2 and VCO2)
Change in blood lactate concentration measured via pinprick capillary blood test | 36, 39 and 42 Days
  Assessed as mmol/L in capillary blood
Change in body composition measured by dual energy X-ray absorptiometry (DXA) | 33 Days
  Assessed as percent fat and muscle mass (%) with a DXA scan
Change in intestinal permeability markers measured in serum | 33 Days
  Assessed in serum as pg/ml (Zonulin, Irisin, and Claudin2)
Change in cytokines | 33 Days
  Assessed in serum as fg/ml (IFN-γ, IL-10, IL-12p70, IL-17, IL-1β, IL-2, IL-4, IL-6, TNF-α)
Change in gastrointestinal symptoms measured by self-report | 33 Days
  Assessed via subjective ratings on a Patient-Reported Outcomes Measurement Information System® (PROMIS®)-GI scale
Change in fecal SCFA concentration measured by gas chromatography | 33 Days
  Assessed as µmol/L of fecal SCFAs (acetate, butyrate, propionate, and total SCFAs)
Synbiotic strains quantification measured by qPCR in fecal matter | 33 Days from Day 0
  Assessed as 16S rRNA gene copies determined with qPCR
Change in fecal microbiota composition | 33 Days
  Assessed as relative abundance of the 16S rRNA amplicon obtained via sequencing
Incidence of adverse events | 42 Days
  Assessed as the number of adverse events and serious adverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: Raylene A Reimer, PhD, RD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada